CLINICAL TRIAL: NCT02348827
Title: Family Psychoeducation for Major Depressive Disorder - a Randomized Controlled Trial
Brief Title: Family Psychoeducation for Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Mental Health Centre North Zealand (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-4-2014-044
Record Dates: First submitted 2015-01-05; First posted 2015-01-28 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Major Depressive Disorder
Keywords: Unipolar depression; Family Therapies; Psychoeducation; Family psychoeducation
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family psychoeducation (Experimental): The intervention consists of group-based family psychoeducation-program aimed at the patients' relatives. Each group will consist of 5 participants and the patients will not be present at group sessions. The program consists of four weekly sessions each consisting of both short lectures on relevant topics as well as interactive séances designed to give participants problem-solving skills.
  Interventions: Behavioral: Family psychoeducation
- Social support group (Active Comparator): Relatives in the social support group will attend the same number of sessions of the same duration, as the relatives in the intervention group (family psychoeducation). The psychiatric nurse who will be in charge of the social support group will not give any psychoeducational intervention.
  Interventions: Behavioral: Social support group

INTERVENTIONS:
Behavioral: Family psychoeducation
  Arms: Family psychoeducation
Behavioral: Social support group
  Arms: Social support group

SUMMARY:
The aim of the present study is to compare an intervention consisting of Family Psychoeducation (FPE) to an active control intervention of social support for relatives of patients with a diagnosis of major depression.

DETAILED DESCRIPTION:
More than 50 % of patients experiencing their first depressive episode will have at least one new episode. Therefore, effective interventions to reduce the risk of relapse are.

Psychoeducation is an interactive education form enhancing knowledge about patients' illness, including it course, symptoms and treatment.

Psychoeducational methods can also act as family intervention which already is an evidence-based practice in schizophrenia and bipolar disorder.

In spite of unipolar depression's high prevalence, only few studies have focused on the effect of psychoeducation, including family psychoeducation, in the prevention of new depressive episodes.

The aim of the present study is to compare an intervention consisting of Family Psychoeducation (FPE) to an active control intervention of social support for relatives of patients with a diagnosis of major depression.

The following hypotheses are proposed:

1. Psychoeducational intervention for relatives will reduces the risk of depressive relapse (defined as a score on The Hamilton six-item subscale, HAM-D6≥7), among remitted depressed patients compared to the control condition
2. Psychoeducational intervention for relatives will shorten time to achieve full symptomatic remission (defined as a score HAM-D6<5) among partially remitted depressed patients compared to the control condition
3. Psychoeducational intervention for relatives will more effectively reduce depressive symptoms (measured on the HAM-D6) among patients fully symptomatic currently depressed patients, compared to control condition.

Secondary aims The study has as a secondary goal to investigate whether a high level of expressed emotion (EE) in relatives at baseline will be associated with poorer outcome, in the form of relapse, in depressed patients.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Age between 18 and 75
* Major depression diagnosis according to the ICD-10 established by a board certified psychiatrist and verified by the MINI International Neuropsychiatric Interview
* Living together , or in very regular contact (every day or almost every day), with an adult relative that the patient considers as emotionally important and who are available for intervention

Regarding hypothesis 1 and 2, patients will be included if they are in remission or partial remission at the inclusion time defined as a score <13 on the Hamilton Rating Scale for Depression (HAM-D17) [20]. Patients included for the test of hypothesis 3 have a HAM-D17-score >13 at the time of the inclusion.

Exclusion Criteria:

* Insufficient knowledge of Danish
* Clinical suspicion of dementia
* Alcohol, drug or medicine abuse
* Psychotic symptoms
* Co-morbidity of severe personality disorder
* Having undergone ECT treatment during the index depressive episode
* Maximum duration of the current depressive episode may not exceed 2 years
* Maximum duration of a period with stable remission may not exceed 3 consecutive months

Regarding to the relatives following criteria for participation apply:

Inclusion criteria:

• Age between 18 and 75

Exclusion criteria:

• Insufficient knowledge of Danish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of relpase | 9 months
  The primary outcome is relapse defined as a score ≥ 7 on HAM-D6 [47] in the 9-month follow-up period (hypothesis 1) among remitted patients.

SECONDARY OUTCOMES:
Time to relapse | Up to 9 months from baseline
  The number of weeks from baseline to relapse, time to full remission defined as a HAM-D6 <5, among the partially remitted patients (hypothesis 2)
Reduction of depressive symptoms | 9 months
  Reduction of depressive symptoms in the HAM-D6-score (hypothesis 3).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Timmerby Timmerby, MD, Principal Investigator — Mental Health Centre North Zealand, Denmark
Locations (1):
- Psychiatric Research Unit, Mental Health Centre North Zealand, Hilleroed, Denmark

REFERENCES:
- [Derived] Timmerby N, Austin SF, Ussing K, Bech P, Csillag C. Family psychoeducation for major depressive disorder - study protocol for a randomized controlled trial. Trials. 2016 Aug 30;17(1):427. doi: 10.1186/s13063-016-1549-0. PMID 27577267
- See also: For information about the project (in Danish) — https://www.psykiatri-regionh.dk/forskning/For-patienter/Sider/psykoedukation_depression.aspx